CLINICAL TRIAL: NCT04217278
Title: An International Randomised Clinical Trial of Therapeutic Interventions to Assess the Effects on Outcome in Adults With Acute Myeloid Leukaemia and High Risk Myelodysplasia Undergoing Allogeneic Stem Cell Transplantation.
Brief Title: A Trial of Treatments to Assess the Effects on Outcome of Adults With AML and MDS Undergoing Allogeneic SCT
Acronym: COSI
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Birmingham (Other)
Collaborators: Jazz Pharmaceuticals (Industry); IMPACT (funded by NHS Blood & Transplant, Anthony Nolan and Leukaemia UK) (Unknown); Adienne SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG_17-234
Record Dates: First submitted 2019-11-20; First posted 2020-01-03 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Acute Myeloid Leukaemia; High-risk Myelodysplastic Syndrome
Keywords: Allogeneic Stem Cell Transplant; AML; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — CPX-351; fludarabine; fludarabine phosphate; Busulfan; Thiotepa; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- R1: Intermediate dose Cytarabine (Active Comparator): First Randomisation (closed to recruitment) - control arm: Intermediate dose Cytarabine (1g/m^2 administered by intravenous infusion over 2 hours on days 1-5 inclusive)
  Interventions: Drug: Cytarabine
- R1: Vyxeos (Experimental): First Randomisation (closed to recruitment) - experimental arm: Vyxeos (29mg/65mg/m^2 administered by intravenous infusion over 90 minutes on days 1 and 3)
  Interventions: Drug: Vyxeos
- R2: FB4 (Active Comparator): Second Randomisation - under 55 years - control arm: Fludarabine (40mg/m^2 days -7, -6, -5, and -4), Busulphan (3.2mg/kg days -7, -6, -5 and -4)
  Interventions: Drug: Fludarabine; Drug: Busulphan
- R2: TBF (Experimental): Second Randomisation - under 55 years - experimental arm: Thiotepa (5mg/kg day -7 and -6), Busulphan (3.2mg/kg days -5, -4 and -3), Fludarabine (50mg/m^2 days -5, -4 and -3)
  Interventions: Drug: Fludarabine; Drug: Busulphan; Drug: Thiotepa
- R3: FB2 (Active Comparator): Third Randomisation - 55 years and over (or under 55 with comorbidities) - control arm: Fludarabine (30mg/m^2 days -6, -5, -4, -3 and -2), Busulphan (3.2mg/kg days -6 and -5)
  Interventions: Drug: Fludarabine; Drug: Busulphan
- Mini-TBF (Experimental): Third Randomisation - 55 years and over (or under 55 with comorbidities) - experimental arm: Thiotepa (5mg/kg day -6), Busulphan (3.2mg/kg days -5 and -4), Fludarabine (50mg/m^2 days -5, -4, and -3)
  Interventions: Drug: Fludarabine; Drug: Busulphan; Drug: Thiotepa

INTERVENTIONS:
Drug: Vyxeos — Vyxeos administered by intravenous infusion
  Other Names: CPX-351
  Arms: R1: Vyxeos
Drug: Fludarabine — Fludarabine administered by intravenous infusion
  Other Names: Fludara
  Arms: Mini-TBF; R2: FB4; R2: TBF; R3: FB2
Drug: Busulphan — Busulphan administered by intravenous infusion
  Other Names: Busulfan; Bulsivex
  Arms: Mini-TBF; R2: FB4; R2: TBF; R3: FB2
Drug: Thiotepa — Thiotepa administered by intravenous infusion
  Other Names: Tepadina
  Arms: Mini-TBF; R2: TBF
Drug: Cytarabine — Cytarabine administered by intravenous infusion
  Other Names: Ara-C; Cytosine arabinoside
  Arms: R1: Intermediate dose Cytarabine

SUMMARY:
Treatment options for older adults with Acute Myeloid Leukaemia (AML) and Myelodysplasia (MDS) are limited. Although stem cell transplantation remains one of the most effective treatments it is associated with severe side effects which have until recently prevented its use in older adults. In the last decade the use of reduced intensity transplants has allowed the extension of the potentially curative effect of transplantation to older patients in whom it was previously precluded. Although a major advance such transplants are associated with a high risk of disease relapse particularly in patients with high risk disease.

This study will evaluate new transplant strategies with the aim of improving the outcome of patients with AML and high risk MDS after stem cell transplantation. Three approaches to improve transplant outcome will be studied:

1. Comparing the new pre-transplant consolidation therapy vyxeos with the standard consolidation therapy (Randomisation 1 is now closed to recruitment).
2. Comparing new conditioning therapies in patients under the age of 55 years
3. Comparing new conditioning therapies in patients aged 55 and over

All patients will be followed up for a minimum of 2 years.

DETAILED DESCRIPTION:
This is a randomised, international, phase II/III, multicentre, clinical trial in patients with AML and MDS undergoing allo-SCT. Patients with AML or MDS who fulfil the eligibility criteria will be invited to participate in the trial across centers performing allo-SCT.

Patients will be randomised to treatment based on a minimisation algorithm prepared at the Cancer Research UK Clinical Trials Unit (CRCTU).

Randomisation 1 (R1) (closed to recruitment) will compare the novel consolidation therapy vyxeos with the standard consolidation therapy intermediate dose cytarabine.

Randomisation 2 (R2) will compare the novel conditioning regimen thiotepa/busulphan/fludarabine (TBF) with the standard conditioning therapy fludarabine/busulphan (FB4) in patients aged under 55 years of age.

Randomisation 3 (R3) will compare the novel conditioning regimen mini thiotepa/busulphan/fludarabine (mini TBF) with the standard regimen fludarabine/busulphan (FB2) in patients aged 55 years of age and over (or patients aged under 55 with comorbidities).

ELIGIBILITY:
Eligibility Criteria for Randomisation 1 (closed to recruitment) Inclusion Criteria for Randomisation 1

1. Patients (≥ 18 years old) with a morphological documented diagnosis of AML or MDS who are deemed fit for allo-SCT with one of the following disease characteristics:

   AML
   * Patients in 1st complete remission (CR1) defined as < 5% blasts
   * Patients in 2nd complete remission (CR2) defined as < 5% blasts
   * Secondary AML (defined as previous history of MDS, antecedent haematological disease or chemotherapy exposure) in CR1 or 2 defined as < 5% blasts MDS
   * Patients with advanced or high risk MDS with an IPSS-R of ≥3.5 (intermediate 3.5 or higher) including intermediate or high risk CMML (e.g. CPSS int-2 or high risk)
2. Patients with an identified HLA identical sibling or suitable matched unrelated donor (suitable match defined as no greater than a single allele mismatch at HLA-A, -B, -C, DQB1 or DRβ1)
3. Patients must be considered suitable/fit to undergo allo-SCT as clinically judged by the Local Investigator
4. Females of and male patients of reproductive potential (i.e., not post-menopausal or surgically sterilised) must use appropriate, highly effective, contraception from the point of commencing therapy until 6 months after treatment
5. Patients have given written informed consent
6. Patients willing and able to comply with scheduled study visits and laboratory tests Exclusion Criteria for Randomisation 1

<!-- -->

1. Patients with contraindications to receiving allo-SCT
2. Female patients who are pregnant or breastfeeding. All women of childbearing potential must have a negative pregnancy test before commencing treatment
3. Adults of reproductive potential not willing to use appropriate, highly effective, contraception during the specified period
4. Patients with renal or hepatic impairment as clinically judged by the Local Investigator
5. Patients with active infection, HIV-positive or chronic active HBV or HCV.
6. Patients with a prior malignancy, except lobular breast carcinoma in situ, fully resected basal cell or squamous cell carcinoma of skin or treated cervical carcinoma in situ, incidental histologic finding of prostate cancer (T1a or T1b using the tumor, node, metastasis (TNM) clinical staging system), previous MDS, CMML, MPN resulting in secondary AML. Cancer treated with curative intent ≥ 5 years previously will be allowed. Cancer treated with curative intent < 5 years previously will not be allowed.
7. History of serious hypersensitivity reaction to cytarabine, daunorubicin, or any component of the Vyxeos formulation.
8. Known history of Wilson's disease or other copper-related metabolic disorder since copper gluconate is a component of the Vyxeos formulation

Eligibility Criteria for Randomisation 2 Inclusion Criteria for Randomisation 2

1. Patients aged between 18 - 54 years with a morphological documented diagnosis of AML or MDS who are deemed fit for a MAC allo-SCT with one of the following disease characteristics: AML o Patients in 1st complete remission (CR1) defined as < 5% blasts

   * Patients in 2nd complete remission (CR2) defined as < 5% blasts
   * Secondary AML (defined as previous history of MDS, antecedent haematological disease or chemotherapy exposure) in CR1 or 2 defined as < 5% blasts
   * Must have received at least two courses of prior intensive chemotherapy prior to transplant unless there are exceptional circumstances. Patients with AML who have achieved CR with Venetoclax based induction regimen treatment as only prior treatment, will also be eligible.

   MDS

   o Patients with advanced or high risk MDS (with an IPSS-R of ≥3.5 (intermediate 3.5 or higher) including intermediate or high risk CMML (e.g. CPSS int-2 or high risk), who have < 10% blasts at the time of randomisation following intensive chemotherapy (including R1 randomisation) or hypomethylating agents if necessary
2. Patients with an identified HLA identical sibling or suitable matched unrelated donor (suitable match defined as no greater than a single allele mismatch at HLA-A, -B, -C, DQB1 or DRβ1)
3. Patients with an ECOG performance status of 0, 1 or 2
4. Patients considered suitable/fit to undergo a MAC allo-SCT as clinically judged by the Local Investigator including:

   1. Adequate hepatic and renal function as determined by full blood count and biochemistry assessment
   2. Resolution of any toxic effects of prior therapy (including radiotherapy, chemotherapy or surgical procedures)
   3. Performance of cardiac or pulmonary function tests (where there is a previous history of cardiac or pulmonary impairment)
5. Females of and male patients of reproductive potential (i.e., not post-menopausal or surgically sterilised) must use appropriate, highly effective, contraception from the point of commencing therapy until 12 months after treatment
6. Patients have given written informed consent
7. Patients willing and able to comply with scheduled study visits and laboratory tests Exclusion Criteria for Randomisation 2

1. Patients with contraindications to receiving a MAC allo-SCT 2. Female patients who are pregnant or breastfeeding. All women of childbearing potential must have a negative pregnancy test before commencing treatment 3. Adults of reproductive potential not willing to use appropriate, effective, contraception during the specified period 4. Patients with renal or hepatic impairment as clinically judged by the Local Investigator 5. Patients with active infection, HIV-positive or chronic active HBV or HCV 6. Patients with a prior malignancy, except lobular breast carcinoma in situ, fully resected basal cell or squamous cell carcinoma of skin or treated cervical carcinoma in situ, incidental histologic finding of prostate cancer (T1a or T1b using the tumor, node, metastasis (TNM) clinical staging system), previous MDS, CMML, MPN resulting in secondary AML. Cancer treated with curative intent ≥ 5 years previously will be allowed. Cancer treated with curative intent < 5 years previously will not be allowed.

Eligibility Criteria for Randomisation 3 Inclusion Criteria for Randomisation 3 1. 1. Patients aged between 55 years or older with a morphological documented diagnosis of AML or MDS who are deemed fit for a RIC allo-SCT (or under the age of 55 with comorbidities which are deemed by the local investigator to preclude safe delivery of a MAC allo-SCT may be considered per investigators discretion) with one of the following disease characteristics: AML

* Patients in 1st complete remission (CR1) defined as < 5% blasts
* Patients in 2nd complete remission (CR2) defined as < 5% blasts
* Secondary AML (defined as previous history of MDS, antecedent haematological disease or chemotherapy exposure) in CR1 or 2 defined as < 5% blasts
* Must have received at least two courses of prior intensive chemotherapy prior to transplant unless there are exceptional circumstances. Patients with AML who have achieved CR with Venetoclax based induction regimen treatment, as only prior treatment, will also be eligible.

MDS

* Patients with advanced or high risk MDS (with an IPSS-R of ≥3.5 (intermediate 3.5 or higher) including intermediate or high risk CMML (e.g. CPSS int-2 or high rsk), who have < 10% blasts at the time of randomisation following intensive chemotherapy (including R1 randomisation) or hypomethylating agents if necessary 2. Patients with an identified HLA identical sibling or suitable matched unrelated donor (suitable match defined as no greater than a single allele mismatch at HLA-A, -B, -C, DQB1 or DRβ1) 3. Patients with an ECOG performance status of 0, 1 or 2 4. Patients considered suitable/fit to undergo a RIC allo-SCT as clinically judged by the Local Investigator including: a. Adequate hepatic and renal function as determined by full blood count and biochemistry assessment b. Resolution of any toxic effects of prior therapy (including radiotherapy, chemotherapy or surgical procedures) c. Performance of cardiac or pulmonary function tests (where there is a previous history of cardiac or pulmonary impairment 5. Females of and male patients of reproductive potential (i.e., not post-menopausal or surgically sterilised) must use appropriate, highly effective, contraception from the point of commencing therapy until 12 months after treatment 6. Patients have given written informed consent 7. Patients willing and able to comply with scheduled study visits and laboratory tests Exclusion Criteria for Randomisation 3

  1. Patients with contraindications to receiving a RIC allo-SCT
  2. Female patients who are pregnant or breastfeeding. All women of childbearing potential must have a negative pregnancy test before commencing treatment
  3. Adults of reproductive potential not willing to use appropriate, effective, contraception during the specified period
  4. Patients with renal or hepatic impairment as clinically judged by the Local Investigator
  5. Patients with active infection, HIV-positive or chronic active HBV or HCV
  6. Patients with a prior malignancies, except lobular breast carcinoma in situ, fully resected basal cell or squamous cell carcinoma of skin or treated cervical carcinoma in situ, incidental histologic finding of prostate cancer (T1a or T1b using the tumor, node, metastasis (TNM) clinical staging system), previous MDS, CMML, MPN resulting in secondary AML. Cancer treated with curative intent ≥ 5 years previously will be allowed. Cancer treated with curative intent < 5 years previously will not be allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival (all randomisations) | 12 and 24 months
  Defined as time from entering the relevant randomisation to the relevant question until death from any cause. Patients who are alive at the end of the trial or have been lost to follow up will be censored at their date last seen. For randomisations 2 and 3 this outcome will also be calculated as time from transplantation in order to run a sensitivity analysis.

SECONDARY OUTCOMES:
Change in MRD status - R1 only | Assessed at baseline and pre-transplant
  Change in minimal residual disease status. A patient will be categorised as either MRD status reduction (MRD positive to negative), MRD remain negative, MRD remain positive or MRD progression (MRD negative to positive) - Randomisation 1 only
Disease-free survival | From date of randomisation through to study completion, an average of 6 years
  DFS defined as time from randomisation to the relevant question to the first of relapse or death from any cause. Patients who are alive and disease free at the end of the trial will be censored at their date known to be alive.
Cumulative incidence of disease relapse | From date of randomisation through to study completion, an average of 6 years
  CIR defined as time from randomisation to the relevant question to the date of relapse. Patients who die prior to relapse will be treated as a competing risk and patients who are alive and relapse free at the end of the trial will be censored at their date last seen.
Non-relapse mortality | From date of randomisation through to study completion, an average of 6 years
  NRM defined as the time from randomisation to the relevant question to date of non-relapse death. Patients who die post-relapse will be treated as a competing risk and patients who are alive at the end of the trial will be censored at their date last seen.
Quality of Life measured by EORTC-QLQ-C30 questionnaires, recorded at multiple timepoints - R2 and R3 only | Assessed at pre transplant, day 28 and months 3, 6, 9, 12, 18 and 24
  The EORTC QLQ-C30 uses for the questions 1 to 28 a 4-point scale. The scale scores from 1 to 4 ("Not at all" to "Very much"). For the raw score, less points are considered to have a better outcome. For the questions 29 and 30 it uses a 7-points scale. The scale scores from 1 to 7 ("very poor" to "excellent"). More points are considered to have a better outcome.
Quality of Life measured by EQ-5D questionnaires, recorded at multiple timepoints - R2 and R3 only | Assessed at pre transplant, day 28 and months 3, 6, 9, 12, 18 and 24
  EQ5D is one of the most widely used health states descriptive system. EQ-5D questionnaires have 5 dimensions: "Mobility", "Human Autonomy," "Current Activities", "Pain / Discomfort", "Anxiety / Depression" and all dimensions are described by 3 problem levels corresponding to patient response choices. A quality of life score is obtained according to the answers to the questionnaires.
Incidence of acute and chronic Graft versus Host Disease - R2 and R3 only | From date of randomisation through to study completion, an average of 6 years
  Incidence of acute and chronic GvHD of any grade - Randomisation 2 and 3 only
Incidence of primary graft failure - R2 and R3 only | From date of randomisation through to study completion, an average of 6 years
  Defined as loss of donor cells after transplantation - Randomisation 2 and 3 only
Incidence of toxicities reported as per CTCAE V4.0 | From start of treatment until 28 days after last dose of treatment
  Defined as the number of patients who report one or more adverse event of grade 3 or higher or a serious adverse event of any grade

CONTACTS AND LOCATIONS:
Overall Officials: Charles Craddock, Professor, Principal Investigator — University Hospital Birmingham NHS Foundation Trust
Locations (14):
- United Kingdom (14):
  - Queen Elizabeth Hospital, Birmingham
  - University Hospitals Bristol, Bristol
  - Addenbrooke's Hospital, Cambridge
  - University Hospital of Wales, Cardiff
  - Queen Elizabeth Hospital Glasgow, Glasgow
  - St James' University Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - Hammersmith Hospital, London
  - King's College Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Freeman Hospital, Newcastle
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: No